CLINICAL TRIAL: NCT02175043
Title: Clinical Benefits of Additional Complex Fractionated Atrial Electrogram Targeted Catheter Ablation for Longstanding Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2014-0282
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, catheter ablation, recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the operation to add in CFAE to conventional liner ablation (Experimental): The group of positive control is the operation to add in CFAE to conventional liner ablation in persistent atrial fibrillation patients
  Interventions: Procedure: atrial electrogram and liner ablation
- only doing conventional liner ablation (Active Comparator): The group of negative is the operation to only doing conventional liner ablation with persistent atrial fibrillation
  Interventions: Procedure: atrial electrogram and liner ablation

INTERVENTIONS:
Procedure: atrial electrogram and liner ablation — 1. The group of positive control is the operation to add in CFAE to conventional liner ablation in persistent atrial fibrillation patients
  2. The group of negative is the operation to only doing conventional liner ablation with persistent atrial fibrillation

SUMMARY:
1. Purpose of the study

1) To compare clinical outcome, procedure time, complication rate of persistent atrial fibrillation patients between conventional additional linear ablation and additional complex fractionated atrial electrogram targeted catheter ablation.

2. Scientific evidence of the study

1. In atrial fibrillation patients, the maintenance of normal sinus rhythm showed significant reduction of mortality.
2. drug therapy with anti-arrhythmic drug showed many complications and side effect, thus non-drug therapy such as catheter ablation is developed.
3. catheter ablation has been performed for 10years world-wide, and showed superior treatment outcome compared with drug therapy.
4. However, there are no consensus for proper ablation strategy in longstanding persistent atrial fibrillation.
5. additional ablation make extent of myocardial injury and paradoxically increase recurrence rate, thus still controversial.
6. Therefore, we will compare conventional linear ablation with additional complex fractionated atrial electrogram targeted catheter ablation.

3. Methods

1. Treatment of All patients with atrial fibrillation is performed according to the standard treatment guideline of atrial fibrillation.
2. there is no additional blood sampling, imaging study, or any other invasive procedure according to the inclusion of the study.

4. study contents

1. to evaluate superior ablation strategy in longstanding persistent atrial fibrillation

   * compare conventional linear ablation with additional complex fractionated atrial electrogram targeted catheter ablation. both strategies are conventional ablation strategies being performed world-wide.
2. compare complex fractionated atrial electrogram before and after linear ablation.

ELIGIBILITY:
Inclusion Criteria:

1) patients who undergoing catheter ablation of atrial fibrillation due to symptomatic, drug refractory atrial fibrillation

Exclusion Criteria:

1. patients who do not agree with study inclusion
2. permanent AF refractory to electrical cardioversion
3. AF with valvular disease ≥ grade 2
4. Patients with left atrial diameter greater than 60mm
5. patients with age less than 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
number of Clinical recurrence of atrial fibrillation (AF) after catheter ablation | 1 year
  lifelong, checked per every outpatient clinic visit

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea